CLINICAL TRIAL: NCT02790658
Title: Metabolomics Approach After Acute Intake of Grumixama Juice (Eugenia Brasiliensis Lam)
Brief Title: Metabolomics Approach After Acute Intake of Grumixama Juice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Luciane de Lira Teixeira, Principal Investigator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 17449613.8.0000.0067
Record Dates: First submitted 2016-04-02; First posted 2016-06-06 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Grumixama; Urolithins; Anthocyanins; Metabolomic Approach; Ellagitannins; Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Grumixama Juice (Other): Juice of grumixama purple fruit (Eugenia brasiliensis Lam.), which is good source of anthocyanins and ellagitannins. It was made with filtered water and sanitized fruits, with a blender. It was administered in single dose of 0.97 mg of anthocyanins and of 4.71 mg of ellagitannins per mL of juice. Which volunteers ingested 10 mL of juice per each Kg body weight.
  The metabolomic approach of plasma and urine samples following acute intake of grumixama juice was done by the collection of blood samples and urine, following the intake of grumixama juice.
  Interventions: Dietary Supplement: Intake of grumixama juice

INTERVENTIONS:
Dietary Supplement: Intake of grumixama juice — In the morning of experimental day after 10 h fasting, the volunteers have been collect the first urine in the morning and it was collected the blood before the intake of grumixama juice, after they drink the juice (0 min), it was collected blood at the times: 15 min, 30 min, 60 min,120 min, 240 min and 24 h; and it was also collected urine at the period: 0 -1h, 1 - 2h, 2 - 4h, 4 - 6 h, 6 - 12 h, 12 - 14 h, the first urine in the morning in the second day (24 h). During the period in the first 4 h of experiment the volunteers only intake the juice.

SUMMARY:
Investigate the bioavailability of the main flavonoid, their colonic transformation and untargeted metabolites by an metabolomic approach following acute intake of a grumixama juice by humans.

DETAILED DESCRIPTION:
The grumixama is a sweet and little cherry native of the South and Southeast regions of the Atlantic Forest of Brazil rich in phenolic compounds, mainly anthocyanins and ellagitannins. The objective of this study is Investigate the bioavailability of the main flavonoid, their colonic transformation and untargeted metabolites by an metabolomic approach following acute intake of a grumixama juice by humans.

Fifteen healthy subjects consumed grumixama juice at single dose, and urine and plasma samples were collected at different time points over 24 h period. The metabolites were analyzed by LC-ESI-MSn, LC-Q-TOF plasma and urine were also analyzed using untargeted metabolomic approach for amino acids and organic acids by GCMS.

ELIGIBILITY:
Inclusion Criteria:

* Not have medical historical of cardiovascular, gastrointestinal, hepatic, renal, thyroid and/or diabetes dysfunction
* Not be alcohol addicts, not use vitamins and other supplements
* Not are using any kind of medication which affect the digestion and absorption of food, not be smokers
* Not are pregnant.

Exclusion Criteria:

* Have medical historical of cardiovascular, gastrointestinal, hepatic, renal, thyroid and/or diabetes dysfunction
* Be alcohol addicts, use vitamins and other supplements
* Are using any kind of medication which affect the digestion and absorption of food, be smokers
* Are pregnant.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2014-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Identification of metabolites in plasma and urine samples of 15 healthy volunteers after intake of grumixama juice by LCMS | 2 months
  The blood and urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins and ellagitannins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by LC-ESI-MSn (for phenolic acids and anthocyanins) and LC-Q-TOF (for urolithins), the mass fragments were expressed in m/z.
Identification of metabolites in plasma and urine samples of 15 healthy volunteers after intake of grumixama juice by GCMS. | 2 months
  The samples were collected as describe in "Arms and Interventions", but for urine samples were used only the samples collected at times 0 (before the juice intake), 0-1h, 1-2h, 2-4h and at 24h after intake. The plasma samples had their proteins precipitated with cold methanol, the metabolites were extracted, concentrated and the amino acids and organic acids were derivatized to became volatile and the samples were analyzed by GCMS. For urine samples the procedures were similar. The mass fragment profile of derivatized compounds were compared to a GCMS library.

SECONDARY OUTCOMES:
Urinary creatinine values of 15 healthy volunteers for data normalization | 15 days
  The creatinine was measured in the 15 volunteers by using a commercial kit, the results obtained in mg/dL, and these values were transformed in mol/L. The values of creatinine were used to normalize the quantification data.
Cycle cell analysis in breast cancer cells treated with metabolites extracted from plasma and urine of 10 healthy volunteers after grumixama juice intake | 2 days
  Plasma and urine preparations were obtained by SPE extraction were dried and tested against breast cancer cells (MDA-MB 231) MDA-MB 231 cells were cultured in monolayer on Dulbecco Eagle modified culture medium supplemented with 10% fetal bovine serum, it was used 5x10-4 cells per well. The cells were incubated in a humidified chamber including 5% CO2 at 37ºC into a confluence of approximately 80%. Cells were further exposed to 200 mg/mL of urine and plasma extract preparations and phenolic compound standards (PCA, VA, HA, C3G) at 0.25 and 25 mg/mL, and maintained at 37ºC, under an atmosphere of 5% CO2 for 48 hours. Negative control was supplied with growth media and DMSO, and blank wells containing growth media only.
  The cells were lysed, the RNA were degraded and the DNA were marked with propidium iodide (1mg/mL) and the fluorescence was measure by flow cytometer and the cell cycle analysis were done by FlowJo. The results were expressed in % of cell for each cell cycle phase.
Multivariate data analysis of metabolites identified in plasma and urine of 15 healthy volunteers after intake of grumixama juice by GCMS | 2 months
  The peak intensity of each compound identified by GCMS were normalized by using a internal standards (D4-alanine). For urine these data also were normalized by creatinine values to normalize sample volume. Multivariate data analysis were done observe changes in these metabolites (amino acids and organic acids) during the 24h after grumixama juice intake. The data were analyzed by MetaboAnalyst 3.0 (http://www.metaboanalyst.ca/).
Pathway analysis of metabolites identified by GCMS | 1 month
  The samples were collected as describe in "Arms and Interventions", but for urine samples were used only the samples collected at times 0 (before the juice intake), 0-1h, 1-2h, 2-4h and at 24h after intake. The plasma samples had their proteins precipitated with cold methanol, the metabolites were extracted, concentrated and the amino acids and organic acids were derivatized to became volatile and the samples were analyzed by GCMS. For urine samples the procedures were similar. The mass fragment profile of derivatized compounds were compared to a GCMS library.
Identification of anthocyanins in urine samples of 10 healthy volunteers by LCMS. | 2 months
  The blood and urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by LC-ESI-MSn (for phenolic acids and anthocyanins) the mass fragments were expressed in m/z.
Identification of phenolic acids in plasma and urine samples of 10 healthy volunteers by LCMS | 2 months
  The blood and urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by LC-ESI-MSn (for phenolic acids and anthocyanins) the mass fragments were expressed in m/z.
Identification of urolithins in urine samples of 10 healthy volunteers by LCMS | 2 months
  The urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the ellagitannins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by LC-Q-TOF (for urolithins), the mass fragments were expressed in m/z.
Quantification of anthocyanins in urine samples of 10 healthy volunteers by HPLC | 2 months
  The urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by HPLC, the results were expressed nmol/mol of creatinine for urine samples. It was made to each volunteer, in each point of collection sample.
Quantification of urolithins in urine samples of 10 healthy volunteers by HPLC | 2 months
  The urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the ellagitannins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by HPLC, the results were expressed in mmol/mol of creatinine. It was made to each volunteer, in each point of collection sample.
Antiproliferative activity of metabolites extracted from plasma of 10 healthy volunteers after grumixama juice intake | 2 days
  Plasma preparations were obtained by SPE extraction were dried and tested against breast cancer cells (MDA-MB 231) MDA-MB 231 cells were cultured in monolayer on Dulbecco Eagle modified culture medium supplemented with 10% fetal bovine serum, it was used 5x10-4 cells per well. The cells were incubated in a humidified chamber including 5% CO2 at 37ºC into a confluence of approximately 80%. Cells were further exposed to 200 mg/mL of plasma extract preparations and phenolic compound standards (PCA, VA, HA, C3G) at 0.25 and 25 mg/mL, and maintained at 37ºC, under an atmosphere of 5% CO2 for 48 hours. Negative control was supplied with growth media and DMSO, and blank wells containing growth media only. Cells were marked with CFSE, and fluorescence was measured by flow cytometer. The results were expressed as % of proliferation inhibition.
Antiproliferative activity of metabolites extracted from urine of 10 healthy volunteers after grumixama juice intake | 2 days
  Urine preparations were obtained by SPE extraction were dried and tested against breast cancer cells (MDA-MB 231) MDA-MB 231 cells were cultured in monolayer on Dulbecco Eagle modified culture medium supplemented with 10% fetal bovine serum, it was used 5x10-4 cells per well. The cells were incubated in a humidified chamber including 5% CO2 at 37ºC into a confluence of approximately 80%. Cells were further exposed to 200 mg/mL of urine extract preparations and phenolic compound standards (PCA, VA, HA, C3G) at 0.25 and 25 mg/mL, and maintained at 37ºC, under an atmosphere of 5% CO2 for 48 hours. Negative control was supplied with growth media and DMSO, and blank wells containing growth media only. Cells were marked with CFSE, and fluorescence was measured by flow cytometer. The results were expressed as % of proliferation inhibition
Quantification of amino acids identified by GCMS | 1 month
  Standards curves of the amino acids that changed significantly after grumixama juice intake were made by GCMS. Through these standards curves the amino acids and organic acids were quantified and the results were expressed in mmol/μmol of creatinine for urine samples and mmol/mL of plasma.
Quantification of organic acids identified by GCMS | 1 month
  Standards curves of organic acids that changed significantly after grumixama juice intake were made by GCMS. Through these standards curves the organic acids were quantified and the results were expressed in mmol/μmol of creatinine for urine samples and mmol/mL of plasma.
Quantification of phenolic acids in plasma samples of 10 healthy volunteers by HPLC | 2 months
  The blood samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by HPLC, the results were expressed in μmol/mL of plasma. It was made to each volunteer, in each point of collection sample.
Quantification of phenolic acids in urine samples of 10 healthy volunteers by HPLC | 2 months
  The urine samples were collected in the times describe in "Arms and Interventions". The samples were acidified and the anthocyanins metabolites were extracted by SPE column, these metabolites extracted were concentrated and analyzed by HPLC, the results were expressed in mmol/mol of creatinine for urine samples. It was made to each volunteer, in each point of collection sample.
Pharmacokinetic parameters (AUC) of anthocyanins in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  Using the quantification results for each collection time was calculated the area under curve (AUC) of anthocyanins in urine (expressed in μmol/h).
Pharmacokinetic parameters (AUC) of phenolic acids in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  Using the quantification results for each collection time was calculated the area under curve (AUC) of phenolic acids in urine (expressed in mmol/h).
Pharmacokinetic parameters (AUC) of urolithins in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  Using the quantification results for each collection time was calculated the area under curve (AUC) of urolithins in urine (expressed in mmol/h).
Urine volume | 1 day
  The volume of each urine sample was measured in mL.
The total elimination of anthocyanins in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  The total elimination amount of anthocyanins was calculated using the urine volume and it was expressed in nmol.
The total elimination of phenolic acids in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  The total elimination amount of phenolic acids was calculated using the urine volume and it was expressed in µmol.
The total elimination of urolithins in urine of 10 healthy volunteers after intake of grumixama juice | 1 month
  The total elimination amount of urolithins was calculated using the urine volume and it was expressed in µmol.

OTHER OUTCOMES:
Normal blood glycemia values of 15 volunteers before juice intake | 1 day
  The glycemia was measured in 15 volunteers to evaluate if the glycemia values were acceptable. The values were expressed in mg/dL.
Normal total cholesterol values of 15 volunteers before juice intake | 1 day
  The total cholesterol was measured in 15 volunteers to evaluate if the cholesterol values were acceptable. The values were expressed in mg/dL.
Normal triglycerides values of 15 volunteers before juice intake | 1 day
  The triglycerides were measured in 15 volunteers to evaluate if the triglycerides values were acceptable. The values were expressed in mg/dL.
Normal HDL values of 15 volunteers before juice intake | 1 day
  The HDL values were measured in 15 volunteers to evaluate if the HDL and LDL values were acceptable. The values were expressed in mg/dL.
Similar weight of 15 volunteers before juice intake | 1 day
  The weight was measured in 15 volunteers to calculate the dose of juice to be give to the volunteers and also to calculate the BMI. The results were expressed in Kg of body mass.
Similar height of 15 volunteers before juice intake | 1 day
  The height was measured in 15 volunteers to calculate the body index mass (BMI). The results were expressed in meters (m).
Similar BMI of 15 volunteers before juice intake | 1 day
  The height was measured in 15 volunteers to calculate the body index mass (BMI). The results were expressed in Kg/m2. This assessment was made to check if the volunteers had a similar BMI.
Normal LDL values of 15 volunteers before juice intake | 1 day
  The LDL values were measured in 15 volunteers to evaluate if the HDL and LDL values were acceptable. The values were expressed in mg/dL.
Normal serum creatinine of 15 volunteers before juice intake | 1 day
  The serum creatinine values were measured in 15 volunteers to evaluate if the values were acceptable. The values were expressed in mg/dL.
Alanine aminotransferase measures in serum samples of 15 volunteers before juice intake | 1 day
  The alanine aminotransferase was measured in the serum of 15 volunteers to evaluate if the values were acceptable. The values were expressed in U/L.
The aspartate transaminase measures in serum samples of 15 volunteers before juice intake | 1 day
  The aspartate transaminase was measured in the serum of 15 volunteers to evaluate if the values were acceptable. The values were expressed in U/L.

CONTACTS AND LOCATIONS:
Overall Officials: Luciane L. Teixeira, MS, Principal Investigator — University of Sao Paulo; Neuza M. Aymoto Hassimotto, PhD, Study Chair — University of Sao Paulo; Franco M. Lajolo, PhD, Study Chair — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flores G, Dastmalchi K, Paulino S, Whalen K, Dabo AJ, Reynertson KA, Foronjy RF, D'Armiento JM, Kennelly EJ. Anthocyanins from Eugenia brasiliensis edible fruits as potential therapeutics for COPD treatment. Food Chem. 2012 Oct 1;134(3):1256-62. doi: 10.1016/j.foodchem.2012.01.086. Epub 2012 Feb 18. PMID 25005941
- [Background] Reynertson KA, Yang H, Jiang B, Basile MJ, Kennelly EJ. Quantitative analysis of antiradical phenolic constituents from fourteen edible Myrtaceae fruits. Food Chem. 2008 Aug 15;109(4):883-890. doi: 10.1016/j.foodchem.2008.01.021. PMID 21340048
- [Background] Teixeira Lde L, Bertoldi FC, Lajolo FM, Hassimotto NM. Identification of Ellagitannins and Flavonoids from Eugenia brasilienses Lam. (Grumixama) by HPLC-ESI-MS/MS. J Agric Food Chem. 2015 Jun 10;63(22):5417-27. doi: 10.1021/acs.jafc.5b01195. Epub 2015 Jun 2. PMID 25990484